CLINICAL TRIAL: NCT07146555
Title: Evaluation of Vitamin D Status in Adult Patients With Newly Diagnosed Immune Thrombocytopenia (ITP)
Brief Title: Vitamin D Satus in Adults With Newly Diagnosed ITP
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Norhan Hassan Mohammed, Resident Doctor in internal Medicine Department at Assiut University hospitals, Assiut University
Other Study IDs: Vitamin D in ITP
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Vitamin D Concentration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected to assess vitamin D level
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First group is responder to ttt of ITP
- 3 groups and assess vitamin D level and its relation with bleeding severity and treatment response
  Interventions: Other: No Interventions
- Second group is non responder to ttt of ITP

INTERVENTIONS:
Other: No Interventions
  Groups: 3 groups and assess vitamin D level and its relation with bleeding severity and treatment response

SUMMARY:
Investigator study aims to assess the level of vitamin D in adult patients with newly diagnosed ITP and correlation between its level and treatment respose

DETAILED DESCRIPTION:
ITP is caused by platelet autoantibodies ,cytotoxic T cell and other factors that accelerate platelet destruction and/or inhibit platelet production . In patients with ITP ,antiplatelet autoantibodies frequently appear to be directed against group Ib /IX and group IIb /IIIa expressed on platelets and megakaryocytes ,both primary and secondary ITP may have an overlapping mechanism of thrombocytopenia and exhibit similar signs and symptoms . The mechanism of ITP associated with other infections e.g (varicella ,HIV, HCV)is at least partly related to molecular mimicry ,Where by antibodies occurring in response to infection subsequently recognize platelet antigens .Abnormalities of cell mediated immunity are known to contribute to pathological process .Like many other autoimmune diseases ,ITP has a T helper cell type 1 bias and a reduced activity of T-regulatory cell.

The role of vitamin D and its prohormones in calcium metabolism and bone formation ,as well as their interaction with immune system , have been the focus of an increasing number of studies in recent years . This is not surprising ,as VD receptors are expressed in a variety of tissues , including the brain ,heart ,skin, bowel gonads ,prostate ,breast and immune cells , in additions to bones , kidneys , and parathyroid . A few autoimmune disorders , including rheumatoid arthritis , and insulin -dependent diabetes mellitus ,have been related to VD deficiency in some recent studies .Based on these association , it has been proposed that VD is an extrinsic factor that can influence the prevalence of autoimmune diseases.

The mechanisms underlaying the link between VD and autoimmunity are not completely identified but probably are related to its anti-inflammatory and immune- modulatory functions. VD appears to interact with immune system through its action on the regulation and differentiation of cells like macrophages ,lymphocytes and natural killer cells in addition to interfering in the in vivo and in vitro production of cytokines .The decrease in the interferon Y- synthesis induced by VD may be one of the methods of VD immune modulatory action . New insights regarding the effect of VD3 derivatives as an immunomodulator .Several studies confirm that VD enhances the innate immune response , Whereas it exercises an inhibitory action on the additive immune system by inhibiting the proliferation of type 1 T- helper cells ,increasing the quantity of type 2 T-helper cells ,increasing the quantity of CD4+/CD25+ T-regulator cells, and inhibiting B cell proliferation , generation of B memory cells ,plasma cell differentiation , and immune globulin production .

The purpose of this study was yo assess the association between adult patients diagnosed with immune thrombocytopenia (ITP) and vitamin D level.

ELIGIBILITY:
Inclusion Criteria:1- Adult (age>18 years) 2-Primary ITP. 3-Patients with ITP who received first line steroid therapy.

Exclusion Criteria:1-Age less than18years 2-Secodary ITP 3-Patients with ITP on second line steroid therapy. 4-Chronic renal disease. 5-Chronic liver disease. 6-Malnutrition and malabsorption.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult patients (>18 years), both male and female, with newly diagnosed immune thrombocytopenia (ITP), recruited from hematology clinics
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Vitamin D Status in Adult Patients with Newly Diagnosed Immune Thrombocytopenia (ITP) | Baseline to 3 months

IPD SHARING:
Plan to Share IPD: Yes